CLINICAL TRIAL: NCT01483430
Title: Effect of Ginseol Kg1 on Blood Pressure Lowering in Prehypertensive or Stage I Hypertensive Patients: Multicenter, Randomized, Placebo-controlled, Double-blind Study
Brief Title: Effect of Ginseol Kg1 on Blood Pressure Lowering
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: DongGuk University (Other)
Responsible Party: Principal Investigator, Kwang-il Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CJ_Ginseol Kg1
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Prehypertension; Hypertension, Stage I
Keywords: Blood pressure; Korea red ginseng; Ambulatory blood pressure; Pulse wave velocity
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ginseol Kg1, high dose (Experimental)
  Interventions: Drug: Ginseol Kg1(high dose)
- Ginseol Kg1, low dose (Experimental)
  Interventions: Drug: Ginseol Kg1 (low dose)

INTERVENTIONS:
Drug: Ginseol Kg1 (low dose) — 1 capsule/day (100mg of Ginseol Kg1), Duration: 8 weeks
  Arms: Ginseol Kg1, low dose
Drug: Ginseol Kg1(high dose) — 1 capsule/day (300mg of Ginseol Kg1), Duration: 8 weeks
  Arms: Ginseol Kg1, high dose
Drug: Placebo — 1 capsule/day (starch), Duration: 8 weeks
  Arms: Placebo

SUMMARY:
In this study, we investigate the effects of Ginseol Kg1 (Korea red ginseng extract) on blood pressure in prehypertensive or stage I hypertensive patients.

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo-controlled, double-blind study. At the end of an initial 2-week washout period, patients fulfilling the inclusion criteria are assigned to three groups, i.e. control group (placebo), low dose Ginseol Kg1 group (100mg), or high dose Ginseol Kg1 (300mg) group. They will intake the study drug for 8 weeks. 24-h ambulatory BP monitoring (ABPM) and pulse wave velocity are measured at the end of the washout period and after 8 weeks of active treatment. At each visit, seated SBP and DBP, heart rate, use of concomitant medication and spontaneously reported adverse events are recorded. Compliance with medication (determined by counting returned tablets) is evaluated at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults over 20 years
* Prehypertension or stage 1 hypertension (systolic blood pressure 120~159mmHg or diastolic blood pressure 80~99mmHg)
* Subject who has not taken medications to treat hypertension within 15 days prior to first visit

Exclusion Criteria:

* Subject who has been involved in other clinical trials within 30 days prior to first visit
* Subject who has following diseases within 2 years prior to screening: angina pectoris, myocardial infarction, heart failure, peripheral vascular disease, chronic liver failure, chronic renal failure, diabetes mellitus, hyperthyroidism, hypothyroidism, malignant tumor, mental disease
* Systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 100 mmHg during screening period
* Subject who has hepatic dysfunction(AST, ALT ≥ 2.5 times higher than normal value)
* Subject who has renal dysfunction(creatinine ≥ 1.5 times higher than normal value)
* Subject who is pregnant or breast feeding
* Alcoholic
* Subject who has an allergy to the ingredients of study product

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The difference of the changes in office diastolic and systolic BP after 8 weeks' treatment between placebo and Ginseol Kg1 group | baseline and 8 week

SECONDARY OUTCOMES:
The difference of the changes in the mean 24-hour ambulatory systolic and diastolic BP after 8 weeks' treatment between placebo and Ginseol Kg1 group. | baseline and 8 week
The difference of the change in the brachial-ankle pulse wave velocity after 8 weeks' treatment between placebo and Ginseol Kg1 group. | baseline and 8 week
The difference of the change in the hs-CRP after 8 weeks' treatment between placebo and Ginseol Kg1 group. | baseline and 8 week
The difference of the change in the lipid profiles after 8 weeks' treatment between placebo and Ginseol Kg1 group | baseline and 8 week
The difference of the changes in office diastolic and systolic BP after 4 weeks' treatment between placebo and Ginseol Kg1 group. | baseline and 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-il Kim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Rhee MY, Cho B, Kim KI, Kim J, Kim MK, Lee EK, Kim HJ, Kim CH. Blood pressure lowering effect of Korea ginseng derived ginseol K-g1. Am J Chin Med. 2014;42(3):605-18. doi: 10.1142/S0192415X14500396. PMID 24871654